CLINICAL TRIAL: NCT05534373
Title: Comparative STudy of the ARGos Biometer Compared to UltraSound Biometer in B-mode in Case of Measure Failure With a the Conventional Biometer
Acronym: STARGUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220627
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-09

CONDITIONS: Cataract
Keywords: ARGOS biometer; UltraSound biometer; conventional biometer; cataract surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Biometry has become one of the most important steps in modern cataract surgery. The axial length of the eye may be measured by ultrasound (either contact or immersion) or by optical means.

Non-contact optical biometry has become the gold-standard because of its ease of use, accuracy, and reproducibility. However, the main disadvantage of the optical methods is their inability to obtain axial length measurements in approximately 10% of eyes, typically those with dense posterior subcapsular cataracts.

By Using SS-OCT device, it has been reported that the AL measurements cannot be made in 0.6 to 7.4% of cases . Therefore, measurement by US biometer is still necessary for advanced cataract. The ultrasound measure the LA between the corneal epithelium and the vitreomacular interface. Ultrasound in B mode (or Brilliance) with the help of the control vector allows a 2-dimensional control of the plan used for measurement. This method is used in current practice in our centers when LA measurements is not possible with our optical SS-biometer.

Recently Alcon has integrated the ARGOS® biometer's diagnostic testing with Alcon's Cataract Refractive Suite technologies. ARGOS® is a non-invasive, non-contact biometer based on swept-source optical coherence tomography (SS-OCT). The device is intended to acquire ocular measurements as well as perform calculations to determine the appropriate intraocular lens (IOL) power and type for implantation during intraocular lens placement. ARGOS® measures the following 9 parameters: Axial Length, Corneal Thickness, Anterior Chamber Depth, Lens Thickness, K-values (Radii of flattest and steepest meridians), Astigmatism, White-to-White (corneal diameter) and Pupil Size. The Reference Image functionality is intended for use as a preoperative and postoperative image capture tool. ARGOS® includes an operation mode for when the retina is hardly or not visible at all denominated the "Enhanced Retinal Visualization mode" (ERV) that allows, in most cases, visualization of the retina. This signal in the retinal region is enhanced by shifting the coherence function (Argos Users manual).

In a prospective observational study conducted in 2 centers in USA involving 107 eyes, they have evaluated the repeatability and reproducibility of ARGOS® measurements in comparison with IOLMaster®500 and LENSTAR LS 900. They have shown that the AL acquisition rate was higher with ARGOS® (96%) compared with both LENSTAR LS 900 (79%) and IOLMaster®500 (77%). The reason was that ARGOS® was more successful at measuring AL in eyes with dense cataract.

DETAILED DESCRIPTION:
Our recent experience with Argos has shown that LA measurements were even possible with our without ERV mode in case of very dense (ie: cataracts in diabetic patients) or posterior subcapsular cataracts.

These observations lead us to propose a retrospective study to compare Argos to our gold standard "ultrasound biometer in mode B" for LA measurements in case of failure with the conventional optical biometer used in our current practice (Lenstar LS900, IOLMaster 500, 700) In current practice, the biometry measurements are conducted with our conventional optical biometer during the visit prior to cataract surgery.

At the same time, measures will be conducted on Argos with or without the ERV mode If axial length measurements are impossible with our conventional optical biometer due to the level of cataract density, axial length measurements will be conducted with our ultrasound biometer in mode-B (Quantel Medical, Aviso S with the 10MHz probe) according to our current practice.

We will retrospectively collect the consecutive data from eyes for which axial length measurements with our conventional biometer were not possible

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* All consecutive patient measured on Argos and any other conventional optical biometer and presenting a failure with one of the conventional optical biometer in AL measurement due to cataract density

Exclusion Criteria:

* Silicon tamponade in the posterior segment
* Patients who are informed and objected to participating to the research
* Patient subject to legal protection measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective observational multicentre non-interventional study including patients whose measurements were performed between August 2021 and January 2022.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
To describe axial length (AL) measured by the Argos biometer in case of measure failure with a conventional optical biometer and to compare it with the AL measured with ultrasound biometry in B-mode (considered to be the gold standard) | 2 months
  Axial length (AL) in millimeters obtained with Argos and ultrasound biometer in B-mode scans (considered to be the reference method for dense cataract)

SECONDARY OUTCOMES:
to describe Pachymetry in micrometers obtained with Argos biometer, conventional biometer and ultrasound biometer | 2 months
  Pachymetry in micrometers obtained with Argos biometer, conventional biometer and ultrasound biometer
to measure anterior chamber depth in millimeters obtained with Argos biometer, conventional biometer and ultrasound biometer | 2 months
  Anterior chamber depth in millimeters obtained with Argos biometer, conventional biometer and ultrasound biometer
to measure lens thickness obtained with Argos biometer and ultrasound biometer | 2 months
  Lens thickness obtained with Argos biometer and ultrasound biometer

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: No